CLINICAL TRIAL: NCT00013585
Title: Phase II, Placebo-Controlled, Double-Blind Study of the Selegiline Transdermal System (STS) in the Treatment of HIV-Associated Cognitive Impairment
Brief Title: Safety and Effectiveness of the Selegiline "Patch" for Decreased Mental Function in HIV Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Neurologic AIDS Research Consortium (NARC) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A5090; 10075 (Registry Identifier: DAIDS ES); ACTG A5090; AACTG A5090
Record Dates: First submitted 2001-03-22; First posted 2001-08-31 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: Cognition Disorders; HIV Infections
Keywords: Cognitive Disorders; AIDS Dementia Complex; Selegiline; Administration, Cutaneous; Neuroprotective Agents
MeSH Terms: conditions — Cognition Disorders; HIV Infections; Cognitive Dysfunction; AIDS Dementia Complex | interventions — Selegiline

INTERVENTIONS:
Drug: Selegiline hydrochloride

SUMMARY:
A decrease in mental function often occurs in patients with HIV. Antiretroviral (ARV) drugs are used to treat this but are not entirely effective. Some other therapy could play a role. The drug selegiline in its pill form is used to treat Parkinson's disease, a serious brain disorder. It is believed this drug might protect the brain and repair some damage. This study will use this drug in a "patch" form, which has not been approved by the Food and Drug Administration (FDA), to see if it helps with decreased mental function in patients with HIV. The purpose of this study is to evaluate the use of selegiline transdermal system (STS) in the treatment of decreased mental function in patients with HIV.

DETAILED DESCRIPTION:
Cognitive impairment is a common adverse effect of HIV infection that can progress to dementia. ARVs are the only current therapy, but treatment response is frequently unsatisfactory, short lived, or the agents are poorly tolerated in doses adequate for central nervous system (CNS) penetration. An adjunctive therapy that interferes with the cascade of events triggered by the virus is likely to play an important role. Oral selegiline is an approved and marketed drug for the symptomatic treatment of Parkinson's disease. Studies suggest that selegiline has a neuroprotective effect and that it may exert a "rescue effect" on dying and injured neurons. This study proposes to use transdermal selegiline, which may deliver a greater dose level than oral administration, in the treatment of HIV-associated cognitive impairment.

This is a two-step study, with each step lasting 24 weeks. Step 1 is double-blind and Step 2 is open label. At entry, patients are randomly assigned to receive either the STS or placebo. One STS patch will be applied daily at the same time for 24 weeks. Patients are evaluated at the clinic at entry and at Weeks 2, 4, 8, 12, 16, and 24. Cognitive status will be evaluated by performance on a series of neuropsychological assessments. Patients who complete Step 1 may participate in Step 2. Patients on placebo in Step 1 will receive active STS treatment in Step 2. The STS patch is applied once daily for an additional 24 weeks and patients are evaluated at the clinic at Weeks 28, 36, and 48.

ELIGIBILITY:
Note: This trial closed to accrual on 12/15/04. Use of the lower-dose STS was discontinued on 05/31/05. Any patients joining the study after 05/31/05 assigned to the interventional arm or who are currently enrolled in Step 2 will receive the higher-dose STS.

Inclusion Criteria:

* HIV infected
* Stable anti-HIV therapy or no anti-HIV therapy for at least 8 weeks prior to study screening
* AIDS Dementia Complex Stage of greater than 0
* Decreased mental function as shown by tests during screening
* IQ of 70 or greater
* Willing to use acceptable methods of contraception during study and for 3 months following study

Exclusion Criteria:

* Tumor involving a large organ or requiring chemotherapy. Patients with basal cell carcinoma, in situ carcinoma of the cervix, or Kaposi's sarcoma are not excluded.
* Serious mental illness that, in the opinion of the investigator, might interfere with the study
* Reserpine or meperidine within 7 days prior to study entry
* Nefazodone within 14 days prior to study entry
* Monoamine oxidase inhibitor, including selegiline, within 30 days prior to study entry
* Sympathomimetic medications, including over the counter diet and cold (oral or nasal) remedies, within 14 days of study entry
* Decreased blood pressure when standing up
* Uncontrolled high blood pressure
* Active symptomatic AIDS-defining opportunistic infection within 30 days prior to study entry
* Nervous system disorders such as multiple sclerosis, stroke, serious head injury, uncontrolled epilepsy, Tourette's syndrome, Huntington's disease, dementias due to alcohol abuse, vitamin B12 deficiency, or syphilis
* CNS infections or neoplasms including cytomegalovirus (CMV) encephalitis, toxoplasmosis, primary or metastatic CNS lymphoma, progressive multifocal leukoencephalopathy, cryptococcal or other fungal meningitis, tuberculous CNS infection, or untreated neurosyphilis
* Any other condition that, in the investigator's opinion, would interfere with the study
* Certain investigational drugs within 30 days before study entry
* Allergic to selegiline or the STS patch
* Pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Change in cognitive performance Week 24 from screening
frequencies of adverse experiences, abnormal results on laboratory tests, changes over time in laboratory tests and vital signs

SECONDARY OUTCOMES:
Clinical global impression by the investigator comparing selegiline-treated arms with the placebo arm
clinical global impression by the subject comparing selegiline-treated arms with the placebo arm
cognitive domain-specific scores compared between selegiline-treated arms and the placebo arm
neuropsychologic function tests (NPZ-8)
fatigue scale (quality of life)
markers of immune activation and oxidative stress/apoptosis
comparison of selegiline and active metabolite steady-state concentrations at Weeks 4, 12, and 24 to cognitive performance
comparison of selegiline and active metabolite steady-state concentrations at Weeks 4, 12, and 24 to historical data in normal volunteers after 7 days of transdermal selegiline administration
comparison of selegiline and active metabolite steady-state concentrations at Week 4 in subjects on ritonavir-containing protease inhibitor (PI) antiviral regimens, subjects on other PI regimens, and subjects on non-PI-containing antiviral regimens

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Schifitto, M.D., Study Chair — Department of Neurology, University of Rochester Medical Center; Ned Sacktor, M.D., Study Chair — Department of Neurology, Johns Hopkins University Bayview Medical Center; David Simpson, M.D., Study Chair — Department of Clinical Neurophysiology, Mount Sinai School of Medicine
Locations (15):
- United States (15):
  - UCLA CARE Center CRS, Los Angeles, California
  - Ucsd, Avrc Crs, San Diego, California
  - Univ. of Hawaii at Manoa, Leahi Hosp., Honolulu, Hawaii
  - Northwestern University CRS, Chicago, Illinois
  - Cook County Hosp. CORE Ctr., Chicago, Illinois
  - Johns Hopkins Adult AIDS CRS, Baltimore, Maryland
  - Massachusetts General Hospital ACTG CRS, Boston, Massachusetts
  - Washington U CRS, St Louis, Missouri
  - Beth Israel Med. Ctr., ACTU, New York, New York
  - Columbia Univ., HIV Prevention and Treatment Medical Ctr., New York, New York
  - Univ. of Rochester ACTG CRS, Rochester, New York
  - Unc Aids Crs, Chapel Hill, North Carolina
  - Hosp. of the Univ. of Pennsylvania CRS, Philadelphia, Pennsylvania
  - The Miriam Hosp. ACTG CRS, Providence, Rhode Island
  - University of Washington AIDS CRS, Seattle, Washington

REFERENCES:
- [Background] Bell JE. An update on the neuropathology of HIV in the HAART era. Histopathology. 2004 Dec;45(6):549-59. doi: 10.1111/j.1365-2559.2004.02004.x. PMID 15569045
- [Background] Koutsilieri E, Scheller C, ter Meulen V, Riederer P. Monoamine oxidase inhibition and CNS immunodeficiency infection. Neurotoxicology. 2004 Jan;25(1-2):267-70. doi: 10.1016/S0161-813X(03)00105-0. PMID 14697901
- [Background] McArthur JC. HIV dementia: an evolving disease. J Neuroimmunol. 2004 Dec;157(1-2):3-10. doi: 10.1016/j.jneuroim.2004.08.042. PMID 15579274
- [Background] Sacktor N, Schifitto G, McDermott MP, Marder K, McArthur JC, Kieburtz K. Transdermal selegiline in HIV-associated cognitive impairment: pilot, placebo-controlled study. Neurology. 2000 Jan 11;54(1):233-5. doi: 10.1212/wnl.54.1.233. PMID 10636157
- [Background] Schifitto G, Kieburtz K, McDermott MP, McArthur J, Marder K, Sacktor N, Palumbo D, Selnes O, Stern Y, Epstein L, Albert S. Clinical trials in HIV-associated cognitive impairment: cognitive and functional outcomes. Neurology. 2001 Feb 13;56(3):415-8. doi: 10.1212/wnl.56.3.415. PMID 11171916
- [Result] Evans SR, Yeh TM, Sacktor N, Clifford DB, Simpson D, Miller EN, Ellis RJ, Valcour V, Marra CM, Millar L, Schifitto G; AIDS Clinical Trials Group and the Neurologic AIDS Research Consortium. Selegiline transdermal system (STS) for HIV-associated cognitive impairment: open-label report of ACTG 5090. HIV Clin Trials. 2007 Nov-Dec;8(6):437-46. doi: 10.1310/hct0806-437. PMID 18042509
- [Result] Schifitto G, Deng L, Yeh TM, Evans SR, Ernst T, Zhong J, Clifford D. Clinical, laboratory, and neuroimaging characteristics of fatigue in HIV-infected individuals. J Neurovirol. 2011 Feb;17(1):17-25. doi: 10.1007/s13365-010-0010-5. Epub 2010 Dec 23. PMID 21181521